CLINICAL TRIAL: NCT05854771
Title: Effects of Single Bout of Yoga Before vs After Eccentric Exercise on Delayed Onset Muscle Soreness.
Brief Title: Effects Of Yoga Before vs After Eccentric Exercise On Delayed Onset Muscle Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01411 SARA KHAN
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Visual Analog Scale; Exercise; Delayed Onset Muscle Soreness; Yoga; Eccentric exercise; Range Of motion
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single bout of yoga before eccentric exercise group (Active Comparator): Yoga poses will be performed before the eccentric exercise of the four muscles group (elbow flexors and extensors, knee extensors and flexors) for a total time duration of 20-30 minutes. To induce delayed onset muscle soreness the participants will be asked to breathe and hold each yoga pose for 6-8 breaths. The participants will perform 6 sets of 10 repetitions of one repetition maximum eccentric drills of the elbow and knee with 3 minutes rest period between each set.
  Interventions: Other: Single bout of yoga before eccentric exercise
- Single bout of yoga after eccentric exercise group (Active Comparator): Yoga poses will be performed after the eccentric exercise of the four muscles group (elbow flexors and extensors, knee extensors and flexors) for a total time duration of 20-30 minutes. To induce delayed onset muscle soreness the participants will be asked to breathe and hold each yoga pose for 6-8 breaths. The participants will perform 6 sets of 10 repetitions of one repetition maximum eccentric drills of the elbow and knee with 3 minutes rest period between each set.
  Interventions: Other: Single bout of yoga after eccentric exercise

INTERVENTIONS:
Other: Single bout of yoga before eccentric exercise — The participants will perform a single bout of the following 5 yoga poses; Child's pose, Thread the needle pose, Eagle arms, Cow face pose, Hands overhead in wide-legged forward bend before the eccentric exercise designed to induce delayed onset muscle soreness for a total time duration of 20-30 minutes. The participants will be asked to breathe and hold each yoga pose for 6-8 breaths. For induction of delayed onset muscle soreness, one repetition maximum of each participant will be calculated first, and on the basis of one repetition maximum the participants will perform 6 sets of 10 repetitions of the eccentric drills of elbow and knee flexors and extensors with 3 minutes rest period between each set.
  Arms: Single bout of yoga before eccentric exercise group
Other: Single bout of yoga after eccentric exercise — The participants will perform a single bout of the following 5 yoga poses; Child's pose, Thread the needle pose, Eagle arms, Cow face pose, Hands overhead in wide-legged forward bend after the eccentric exercise designed to induce delayed onset muscle soreness for a total time duration of 20-30 minutes. The participants will be asked to breathe and hold each yoga pose for 6-8 breaths. For induction of delayed onset muscle soreness, one repetition of each participant will be calculated first and on the basis of one repetition maximum the participants will perform 6 sets of 10 repetitions of the eccentric drills of elbow and knee flexors and extensors with 3 minutes rest period between each set.
  Arms: Single bout of yoga after eccentric exercise group

SUMMARY:
The goal of this clinical trial is to compare the effects of pre and post-exercise yoga after eccentric exercise on delayed onset muscle soreness in healthy adults. The main question it aims to answer is whether there will be a difference in the effects of pre and post-exercise yoga in reducing delayed muscle soreness. The participants will be divided into two groups; group A and group B. Group A will perform single bout of yoga before the eccentric exercise and Group B will perform single bout of yoga after eccentric exercise.

DETAILED DESCRIPTION:
Delayed onset muscle soreness is a multifactorial well-known phenomenon associated with swelling, tenderness, altered joint kinematics, muscle fiber disruption, acute tissue damage, decreased strength and power, and stiffness. Delayed onset muscle soreness are experienced by both elite and novice athletes after exposure to unaccustomed or strenuous exercise that particularly involves eccentric contractions. The symptoms can range from mild muscle tenderness to severe agonizing pain. According to the "Munich Consensus Statement", Delayed onset muscle soreness is an overexertion-functional muscle disorder that involves type Ib fibers. The intensity of discomfort and soreness associated with delayed onset muscle soreness depends on the level of fitness, type, and repetitions of exercise performed with eccentric exercises resulting in micro injury at a greater frequency and severity in comparison to other exercises. The intensity of delayed onset muscle soreness increases within the first 24 hours and peaks between 24-72 hours. The symptoms of delayed onset muscle soreness subside within 5-7 days after the exercise and thus differ from normal muscle soreness that occurs immediately after the exercise. Although delayed onset muscle soreness is considered a mild type of muscle injury, however; it can affect athletic performance to a great level by causing a reduction in joint range of motion, shock attenuation, and peak torque. Numerous treatment strategies have been used lately to reduce the incidence of delayed onset muscle soreness including hyperbaric oxygen, anti-inflammatory medication, massage, cryotherapy, homeopathy, stretching, electrotherapeutic modalities, ultrasound, rest, light exercise, and yoga. Yoga is a process of physical and mental reconditioning that involves simple meditation, the adoption of certain postures, and breath control. The various health benefits associated with yoga include improved flexibility and balance, muscle strength, skeletal muscle oxygen uptake, lung function, pain relief, and lower stress levels. Depending upon the type, intensity, and the number of repetitions of exercise various yoga poses can be performed before and after eccentric exercises as a warmup or a cool-down procedure to prevent delayed onset muscle soreness.

The current study is aimed to fill the literature gap by finding the difference in the effects of pre and post-exercise yoga poses in reducing delayed onset muscle soreness. This study will provide a guide to elite and novice athletes to effectively incorporate yoga poses in their exercise protocol to prevent delayed onset muscle soreness that results in decreased performance.

ELIGIBILITY:
Inclusion Criteria:

* Untrained men and women
* Aged between 18-30 years
* Body mass index less than 30
* Asymptomatic of disease and illness

Exclusion Criteria:

* Any injury in the arms and/or legs that caused a visit to a medical provider
* Participants who are unable to perform any of the yoga pose.
* High blood pressure
* Pregnant
* Diabetes
* Any nerve, muscle, or joint disorder

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 1 week
  The visual analog scale is used to measure perceived pain which is one of the symptoms of delayed onset muscle soreness. The visual analog scale is a 100-mm continuum with perceived levels of muscle soreness ranging from "No pain" to "Worst possible pain". The score is obtained by measuring the distance in millimeters marked by the respondent from the zero end of the scale. Visual analog scale pain/ soreness scales have been found to be a reliable and valid tool for assessing pain and muscle soreness with an intraclass correlation value (ICC=0.97)
Range of Motion | 1 week
  The range of motion is the measurement of movement around a specific joint or body part. To measure the range of motion, a goniometer is used. A goniometer is a device that measures an angle or permits the rotation of an object to a definite position. The inter-examiner reliability values of goniometer for measuring elbow and knee range of motion ranged from (ICC 0.26-0.96).
Strength | 1 week
  The low-cost digital dynamometer is used to measure the isometric strength of the muscles. The low-cost digital dynamometer has a strong concurrent validity (ICC>0.9) and a high intra and inter-tester reliability (ICC>0.75) for measuring isometric strength of the lower and upper extremity movements.

CONTACTS AND LOCATIONS:
Overall Officials: Jawad Naweed, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Ginnastic Arena, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No